CLINICAL TRIAL: NCT05627193
Title: Comparison of Patient Satisfaction in Post-operative Breast Surgery Patients Having Physical Clinic and Tele Clinic Follow up: A Randomized Controlled Trial (PSPVT Trial)
Brief Title: Comparing Patient Satisfaction in Post-operative Breast Surgery Patients Having Physical Clinic and Tele Clinic Follow up: A Randomized Controlled Trial
Acronym: PSPVT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaukat Khanum Memorial Cancer Hospital & Research Centre (Other)
Responsible Party: Principal Investigator, Dr. Muhammad Awais Kanwal, Principal Investigator, Shaukat Khanum Memorial Cancer Hospital & Research Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB-22-34
Record Dates: First submitted 2022-11-15; First posted 2022-11-25 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Satisfaction, Patient; Satisfaction
Keywords: patient satisfaction; teleclinic; physical clinic; outpatient clinic; breast surgery; virtual clinics; randomized controlled trial; RCT; PSPVT Trial
MeSH Terms: conditions — Patient Satisfaction; Personal Satisfaction | interventions — Ambulatory Care Facilities

STUDY DESIGN:
Intervention Model Description: Pre-operative randomization will be carried out and patients will be allocated to either of the two groups this will be done by 'Computerized block randomization'.
Who Masked: Outcomes Assessor
Masking Description: Assessor determining the patient satisfaction will be blinded to the type of follow up. This will be ensured by restricting the information available to accessor to only the name and contact number of the patient. The assessor will therefore have no access to the electronic health record of the patient on HIS and will not be able to determine the type of follow up of the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional out patient clinic (Active Comparator): The volunteers of the study randomized into this group will be given traditional outpatient clinic follow up post surgery.
  Interventions: Other: Physical Clinic
- Teleclinic (Active Comparator): The Volunteer of the study randomized into this group will be given teleclinic appointment for follow up post surgery.
  Interventions: Other: Teleclinic

INTERVENTIONS:
Other: Teleclinic — Instead of visiting surgeon after travelling from far flung areas for a post surgery follow up appointment, the follow up visit will be done using telephone.
  Other Names: Virtual Clinic; Phone Clinic; Remote Clinic
  Arms: Teleclinic
Other: Physical Clinic — Patients will have to travel to come physically to hospital to meet the operating surgeon.
  Other Names: Traditional Clinic; Outpatient clinic; Standard Clinic
  Arms: Traditional out patient clinic

SUMMARY:
The Purpose of this study is to measure patient satisfaction in standard Post- operative Breast Outpatient clinics versus teleclinics.

Post operative breast surgery patients who volunteer for this study will be randomized into either of the two groups Standard outpatient physical clinics or Telephone clinic and their satisfaction will be measured afterwards using a validated standardized questionnaire by a assessor who will be blind to the type of follow up.

This will be a single blinded randomized controlled trial.

DETAILED DESCRIPTION:
The incidence of Breast Cancer is increasing in Pakistan and worldwide. In 2018, 2.1 million new cases were reported, with 627,000 deaths. Pakistan has the highest incidence of breast cancer among Asian countries: one in nine women is at risk of being diagnosed with breast cancer during their lifetime. According to the International Agency of Research on Cancer 2018 report, 34,066 new cases of breast cancer had been reported in Pakistani women. The Outpatient department Clinics are a standard part of routine follow-up for post-operative patients. Conventional Outpatient clinics incur hefty financial costs on patients living in distant areas.

Access to the telephone is increasing worldwide as technology advances and becomes more accessible to patients. Its use in healthcare settings is inevitable. In post-operative setting, remote consultation is feasible as the usual discussion is about the histopathology report of the procedure performed along with referrals for Adjuvant treatment. Nonetheless, there are some hesitations with this type of consultation. For instance, a visit to a physical clinic may help in early detection of potential complications which may be missed in remote consultation. Similarly, patients may not be satisfied with remote consultation alone.

Tele clinics, which became popular in the wake of Coronavirus disease pandemic, have been instrumental in improving healthcare delivery in Breast Surgery patients and this has been demonstrated by multiple studies but the data regarding patient satisfaction is not available in our population and needs to be studied.

Study Design: Randomized Controlled Trial

Setting: Department of surgical oncology, Shaukat Khanum Memorial Cancer Hospital and Research Centre, Lahore.

Enrolment: Patients will be enrolled pre-operatively, in the holding bay prior to the surgery.

Sample Size: A sample of 182 participants (91 in each group) has been determined for this study. The calculations were based on a 5% level of significance, a 95% confidence interval, 5% margin of error, pooled standard deviation of 3.01, and mean difference of satisfaction score as 1.1 and non-response rate of 5%. Sample size was calculated based on similar research results

Study Duration: Four months after the initiation of enrolment

Follow up Schedule: 2 weeks after surgery, either in physical clinic or tele clinic

Randomization: Pre-operative randomization will be carried out and patients will be allocated to either of the groups by selecting the name of the group to which patient has been randomized from a sealed envelope. The type of randomization would be 'Computerized block randomization'. Research Randomizer software, a free to use software will be used for this.

Blinding: Assessor determining the patient satisfaction will be blinded to the type of follow up. This will be ensured by restricting the information available to accessor to only the name and contact number of the patient. The assessor will therefore have no access to the electronic health record of the patient and will not be able to determine the type of follow up of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Breast Cancer.
* Written informed consent for participation in the trial.

Exclusion Criteria:

* Stage IV Breast Cancer.
* Chronic Pain.
* Breast Surgery with reconstruction.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction | 3 weeks
  Patient satisfaction will be measured using Patient satisfaction questionnaire Short Form (PSQ-18). The short-form instrument, the PSQ-18, contains 18 items tapping each of the seven dimensions of satisfaction with medical care: general satisfaction, technical quality, interpersonal manner, communication, financial aspects, time spent with doctor, and accessibility and convenience. PSQ-18 is a free to use validated tool developed by RAND Corporation.

SECONDARY OUTCOMES:
Post operative complications | 6 weeks
  These will be recorded as per Clavien Dindo Classification (CDC) Grade I Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions Allowed therapeutic regimens are: drugs as antiemetic, antipyretics, analgesics, diuretics and Electrolytes and physiotherapy. This grade also includes wound infections opened at the bedside.
  Grade II Requiring pharmacological treatment with drugs other than such allowed for grade I complications. Blood transfusions and total parenteral nutrition are also included.
  Grade III Requiring surgical, endoscopic or radiological intervention Grade IIIa Intervention not under general anesthesia Grade IIIb Intervention under general anesthesia Grade IV Life-threatening complications (including CNS complications) * requiring IC/ICU-management Grade IVa Single organ dysfunction (including dialysis) Grade IVb Multi-organ Dysfunction Grade V Death of a patient
Number of Emergency assessment room visits prior to follow up in Physical or Tele Clinic | 2 weeks
  If a patient visits Emergency assessment room prior to follow up appointment it will be recorded as it can affect the patient satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Shaukat Khanum memorial cancer hospital and research centre, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with interests in patient satisfaction. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review of a research proposal. for more information PI can be contacted at awaiskanwal@gmail.com

REFERENCES:
- [Background] Khan NH, Duan SF, Wu DD, Ji XY. Better Reporting and Awareness Campaigns Needed for Breast Cancer in Pakistani Women. Cancer Manag Res. 2021 Mar 2;13:2125-2129. doi: 10.2147/CMAR.S270671. eCollection 2021. PMID 33688255
- [Background] McMaster T, Wright T, Mori K, Stelmach W, To H. Current and future use of telemedicine in surgical clinics during and beyond COVID-19: A narrative review. Ann Med Surg (Lond). 2021 Jun;66:102378. doi: 10.1016/j.amsu.2021.102378. Epub 2021 May 8. PMID 33996071
- [Background] Berg WT, Goldstein M, Melnick AP, Rosenwaks Z. Clinical implications of telemedicine for providers and patients. Fertil Steril. 2020 Dec;114(6):1129-1134. doi: 10.1016/j.fertnstert.2020.10.048. PMID 33280717
- [Background] Nomura A, Tanigawa T, Muto T, Oga T, Fukushima Y, Kiyosue A, Miyazaki M, Hida E, Satake K. Clinical Efficacy of Telemedicine Compared to Face-to-Face Clinic Visits for Smoking Cessation: Multicenter Open-Label Randomized Controlled Noninferiority Trial. J Med Internet Res. 2019 Apr 26;21(4):e13520. doi: 10.2196/13520. PMID 30982776
- [Background] Adams L, Lester S, Hoon E, van der Haak H, Proudman C, Hall C, Whittle S, Proudman S, Hill CL. Patient satisfaction and acceptability with telehealth at specialist medical outpatient clinics during the COVID-19 pandemic in Australia. Intern Med J. 2021 Jul;51(7):1028-1037. doi: 10.1111/imj.15205. Epub 2021 Jul 2. PMID 34213046
- [Background] Orrange S, Patel A, Mack WJ, Cassetta J. Patient Satisfaction and Trust in Telemedicine During the COVID-19 Pandemic: Retrospective Observational Study. JMIR Hum Factors. 2021 Apr 22;8(2):e28589. doi: 10.2196/28589. PMID 33822736